CLINICAL TRIAL: NCT01772589
Title: Effect of Cutting Blades for Total Knee Arthroplasty on Implant Migration. A Randomized Controlled Study With Radiostereometric Analysis
Brief Title: Effect of Cutting Blades for Total Knee Arthroplasty on Implant Migration
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Comparator sawblade no longer available
Sponsor: Glen Richardson (Other)
Responsible Party: Sponsor-Investigator, Glen Richardson, MD FRCPC, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: SAW BLD
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- New saw blade (Active Comparator): New saw blade
  Interventions: Procedure: New saw blade
- Reprocessed saw blade (Active Comparator): Reprocessed saw blade
  Interventions: Procedure: Reprocessed saw blade

INTERVENTIONS:
Procedure: New saw blade
  Arms: New saw blade
Procedure: Reprocessed saw blade
  Arms: Reprocessed saw blade

SUMMARY:
There have been considerable efforts to control rising health care costs. One of the more recent developments is the practice of reprocessing single use medical devices. This practice has been shown to provide considerable savings for health care payers. Medical devices have been reprocessed in a number of different medical fields including Orthopaedic Surgery. One of the devices that has been reprocessed are the Precision Saw Blades from Stryker Inc. These saw blades are used during Total Knee Arthroplasty (TKA) surgery. The reprocessed Precision saw blades are Health Canada approved and are available at Capital Health.

Beyond the benefits to the environment and cost savings, the investigators do not know if the reprocessed saw blades work better, work worse or the same as non reprocessed saw blades. This study is designed to determine if the reprocessed saw blades used during a TKA work as well as a new saw blade.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic osteoarthritis of the knee indicating surgical intervention
2. Between the ages of 21 and 80 inclusive
3. Ability to give informed consent

Exclusion Criteria:

1. Significant co-morbidity affecting ability to ambulate
2. Flexion contracture greater than 15°
3. Extension lag greater than 10°
4. Tibial subluxation greater than 10 mm on standing AP radiograph
5. Prior arthroplasty, patellectomy or osteotomy with the affected knee
6. Lateral or medial collateral ligament instability (> 10° varus/valgus)
7. Leg length discrepancy greater than 10 mm
8. Bone quality precluding uncemented fixation
9. Pregnancy
10. Active or prior infection
11. Morbid Obesity (BMI > 40)
12. Medical condition precluding major surgery
13. Severe osteoporosis or osteopenia
14. Neuromuscular impairment

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Implant migration | 2 years
  Implant migration assessed with RSA

SECONDARY OUTCOMES:
Economics | 1 year
  Cost comparison of saw blades

CONTACTS AND LOCATIONS:
Overall Officials: Glen Richardson, MD, Principal Investigator — Capital Health, Canada
Locations (1):
- Capital District Health Authority, Halifax, Nova Scotia, Canada